CLINICAL TRIAL: NCT05407506
Title: Clinical Study of Ultrasonic Artificial Intelligence and Fine Needle Aspiration in Qualitative Diagnosis of Thyroid Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Luo Dingcun (Other)
Responsible Party: Sponsor-Investigator, Luo Dingcun, vice president of hospital, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZhejiangU20220602
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THYROID AI (Experimental)
  Interventions: Diagnostic Test: THYROID AI

INTERVENTIONS:
Diagnostic Test: THYROID AI — thyroid artificial intelligence diagnosis system and fine needle puncture in the diagnosis of benign and malignant thyroid nodules

SUMMARY:
To study the value of thyroid artificial intelligence diagnosis system and fine needle puncture in the diagnosis of benign and malignant thyroid nodules, so as to provide evidence-based medical evidence for the diagnosis of benign and malignant thyroid nodules by artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-75 years old, regardless of gender; (2) The nodules were observed with complete transverse and longitudinal standard sections; (3) The nodules were observed and underwent thyroid fine needle aspiration, including cytology and BRAF gene mutation detection; (4) Patients voluntarily entered the study after informed consent.

Exclusion Criteria:

* (1) If the observed nodule is less than 2mm or more than 50mm, the artificial intelligence system cannot recognize it; (2) Uncontrolled subacute thyroiditis and hyperthyroidism; (3) Previous thyroid surgery or radiofrequency ablation of thyroid nodules; (4) History of neck trauma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
THYROID AI | immediately after the procedure
  classify thyroid nodules as Benign or Malignant

CONTACTS AND LOCATIONS:
Overall Officials: Dingcun Luo, Principal Investigator — First People's Hospital of Hangzhou

IPD SHARING:
Plan to Share IPD: No